CLINICAL TRIAL: NCT05475782
Title: Spyglass-guided Lithotripsy Vs ESWL for Pancreatic Duct Stones
Brief Title: Spyglass-guided Lithotripsy Versus ESWL for Pancreatic Duct Stones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Jianfeng Yang, Professor, First People's Hospital of Hangzhou
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-07-25
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Pancreatic Duct Stone

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spyglass group (Active Comparator): lithotripsy through Spyglass and ERCP
  Interventions: Procedure: Spyglass-guided lithotripsy
- ESWL group (Experimental): Lithotripsy through ESWL and ERCP
  Interventions: Procedure: ESWL

INTERVENTIONS:
Procedure: Spyglass-guided lithotripsy — Spyglass-guided lithotripsy
  Other Names: Direct vision system
  Arms: Spyglass group
Procedure: ESWL — ESWL+ERCP
  Other Names: Lithotripsy through ESWL
  Arms: ESWL group

SUMMARY:
Overall stone clearance with endoscopic retrograde cholangiopancreatography (ERCP) for pancreatic duct stones is a amjor problem, especially bigger size stones. After ERCP failure, surgery was the only option but patients not suitable for surgery were treated through stenting. But had to undergo multiple ERCPs and show lower success rate. Recently, SpyGlass and extracorporeal shock wave lithotripsy (ESWL) have been applied for the treatment of huge stones. The present study aims to compare the efficacy and safety outcomes of SpyGlass-guided lithotripsy and ESWL procedures for the removal of pancreatic duct stones.

DETAILED DESCRIPTION:
ESWL was first used for the removal of renal calculi and ureteral calculi however, now a day is being used for pancreatic duct stones and biliary calculi. It has the advantages of simple operation, lower cost, and higher safety. Recent studies show that the procedure time for ESWL is also shorter and the utilization rate of mechanical lithotripsy was effectively reduced with fewer complications. But It is difficult for ESWL to break the stones larger than 3cm into small pieces.

Spyglass has been used in clinics for more than ten years. Recently, a study reported difficult bile duct stones that were treated with SpyGlass-guided laser lithotripsy that shows promising results. Compared with laser lithotripsy under X-ray monitoring, there is no significant difference in stone removal rate and complication rate between the two methods. However, the effect of lithotripsy under Spyglass direct vision is better, which can break large stones into smaller pieces, thus making it easier to take stones. Investigator conducted the current study to compare the therapeutic outcome and complications between SpyGlass direct vision lithotripsy and ESWL procedures for the removal of large pancreatic duct stones.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic duct sone
* Falied to eliminate through ERCP only

Exclusion Criteria:

* Pregnancy
* Refusal of written informed consent
* Patients not suitable for ESWL/ Spyglass
* Contraindications to ERCP exist
* Complicated with acute pancreatitis or acute cholangitis
* Coagulation dysfunction#thrombocytopenia
* Patients after gastrointestinal reconstruction
* Allergic to drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Technical success | Intraoperative
  Successfull intervention
Clinical success | 1 month
  Pancreatic duct stone clearance rate

SECONDARY OUTCOMES:
Adverse events | 1 month
  procedure related adverse events, bleeding, pancreatitis, etc
Total number of ERCP | 1 month
  Number of ERCPs performed for stone clearnce
Procedure sessions | 1 month
  Total sessions of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Yang, MD, Principal Investigator — Affilated Hangzhou First People Hospital
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guzman-Calderon E, Martinez-Moreno B, Casellas JA, Aparicio JR. Per-oral pancreatoscopy-guided lithotripsy for the endoscopic management of pancreatolithiasis: A systematic review and meta-analysis. J Dig Dis. 2021 Oct;22(10):572-581. doi: 10.1111/1751-2980.13041. PMID 34436824
- [Background] Bick BL, Patel F, Easler JJ, Tong Y, Watkins JL, McHenry L, Lehman G, Fogel EL, Gromski MA, Sherman S. A comparative study between single-operator pancreatoscopy with intraductal lithotripsy and extracorporeal shock wave lithotripsy for the management of large main pancreatic duct stones. Surg Endosc. 2022 May;36(5):3217-3226. doi: 10.1007/s00464-021-08631-7. Epub 2021 Jul 15. PMID 34264399
- [Result] Tandan M, Reddy DN. Extracorporeal shock wave lithotripsy for pancreatic and large common bile duct stones. World J Gastroenterol. 2011 Oct 21;17(39):4365-71. doi: 10.3748/wjg.v17.i39.4365. PMID 22110261
- [Result] van Huijgevoort NCM, Veld JV, Fockens P, Besselink MG, Boermeester MA, Arvanitakis M, van Hooft JE. Success of extracorporeal shock wave lithotripsy and ERCP in symptomatic pancreatic duct stones: a systematic review and meta-analysis. Endosc Int Open. 2020 Aug;8(8):E1070-E1085. doi: 10.1055/a-1171-1322. Epub 2020 Jul 21. PMID 32743061
- [Result] Beyna T, Neuhaus H, Gerges C. Endoscopic treatment of pancreatic duct stones under direct vision: Revolution or resignation? Systematic review. Dig Endosc. 2018 Jan;30(1):29-37. doi: 10.1111/den.12909. Epub 2017 Jul 27. PMID 28656688